CLINICAL TRIAL: NCT06340750
Title: A Phase I Study of BAFF CAR-T Cells (LMY-920) for Treatment of Systemic Lupus Erythematosus
Brief Title: BAFF CAR-T Cells (LMY-920) for Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luminary Therapeutics (Industry)
Collaborators: Nationwide Children (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LMY-920-003
Record Dates: First submitted 2024-03-12; First posted 2024-04-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BAFF CAR T (Experimental): Autologous BAFF CAR T Therapy
  Interventions: Biological: LMY-920

INTERVENTIONS:
Biological: LMY-920 — CAR T Therapy
  Other Names: BAFF CAR T

SUMMARY:
This phase 1 study seeks to examine the safety and recommended phase 2 dose (RP2D) of BAFF-ligand CAR-T cells (LMY-920) in adult patients with refractory systemic lupus erythematosus (SLE). It is hypothesized that BAFF CAR-T cells will be safe and will improve SLE disease activity scores.

DETAILED DESCRIPTION:
This is an open label, phase 1 dose escalation study designed to establish the safety and RP2D of autologous BAFF CAR-T cells in adults with refractory SLE. The planned dose escalation includes 3 dose levels and one de-escalation level. The maximum tolerated dose (MTD) will be determined using a 3+3 dose escalation design. The MTD dose level cohort may be expanded to a total of 6 patients. RP2D may be selected at dose level(s) at or below the MTD based on all data then available (e.g. efficacy, safety, PK and PD), and additional patients enrolled at these levels to expand up to a total of 40 patients in the study, in order to further evaluate safety and efficacy and guide Phase 2 trial design.

To ensure patient safety, during dose escalation, treatment of subjects at each dose will be staggered by at least 14 days. For example, the second subject will be enrolled only after the first subject has finished 14 days of safety monitoring from the CAR-T cell infusion, and the third subject will be enrolled only after the second subject has finished 14 days of safety monitoring from the CAR-T cell infusion. In the expansion cohorts, this staggering interval will no longer be required.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years
* Confirmed Systemic Lupus Erythematosus (SLE) as per Systemic Lupus International Collaborating Clinics (SLICC) 2012 Criteria with one or more of the following:

  a. Active disease despite use of standard therapy (i) and one or more additional therapies (ii).

  i. Corticosteroids (CS), Hydroxychloroquine ii. Mycophenolate mofetil (MMF), Methotrexate (MTX), Azathioprine (AZA), Tacrolimus (TAC), Cyclophosphamide (CYC), Rituximab, and/or belimumab b. Active disease due to intolerance of standard therapy (i) and one or more additional therapies (ii).

  c. Steroid-Dependent Disease
* Subjects must meet organ function criteria:

  1. Creatinine clearance more than or equal to 30 ml/min calculated by the Cockcroft - Gault formula
  2. Subjects must have adequate cardiac function as defined as left ventricular ejection fraction ≥ 40% on the most recent echocardiogram.
  3. Adequate pulmonary function with pulse oximetry ≥92% on room air
  4. Total Bilirubin ≤ 1.5x the institutional upper limit of normal (except in patients with Gilbert's syndrome)
  5. ALT (SGPT) and AST (SGOT) < 3x the institutional upper limit of normal

Exclusion Criteria:

* SLE complicated by:

  * Active neuropsychiatric lupus
  * Active secondary hemophagocytic lymphohistiocytosis (sHLH)
* Presence of any medical or psychological conditions which may affect patient ability to comply with study protocol requirements and study visits
* Presence of active, untreated infection such as:

  * Active microbial infection. Patients with possible fungal infections must have had at least 2 weeks of appropriate anti-fungal therapy and be asymptomatic. Patients with active tuberculosis must have had at least 4 weeks of appropriate anti-mycobacterial treatment and be asymptomatic.
  * Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening
  * HIV positive test within 8 weeks of screening
* Acute/ongoing neurologic toxicity > Grade 1 except for a history of controlled seizures or fixed neurologic deficits that have been stable/improving over the past 1 months.
* Patients with concomitant genetic syndrome: such as patients with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Patients with Down Syndrome will not be excluded.
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study. Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 6 months after the CAR-T cell infusion.
* A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Men who will not agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm, as defined below:
* With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the CAR-T cell infusion. Men must refrain from donating sperm during this same period.
* With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the CAR- T cell infusion to avoid potential embryonal or fetal exposure. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Patients receiving a live vaccines within the last two weeks.
* A minimum of 28 days must have elapsed between prior treatment with investigational agent(s) and the day of lymphocyte collection.
* Concurrent use of high dose systemic steroids and/or T cell directed immune suppression. Subjects must discontinue T cell targeted therapy >3 weeks and wean prednisone dose to ≤10 mg/day prior to leukapheresis.
* Previous treatment with any gene or adoptive cell therapy products.
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, serious arrhythmia, HIV, seizure disorder, cerebrovascular disease, psychiatric disease), that may interfere with the patient's ability to tolerate the therapy or comply with assessments.
* Active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast). Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial (e.g. Low Gleason score prostate Cancer).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Safety of the Treatment | 5 years
  The rate of adverse events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (National Cancer Institute) and rate of dose limiting toxicities after treatment with autologous BAFF CAR-T cells in adults with refractory SLE
Recommended Phase 2 Dose (RP2D) | 5 years
  A dose of autologous BAFF CAR-T cells in adults with refractory SLE less than or equal to that at which less than or equal to 1/6 patients experience dose limiting toxicities.

SECONDARY OUTCOMES:
Efficacy of the Treatment: SELENA-SLEDAI | 5 years
  The change between baseline and post BAFF CAR-T cell infusion SLE disease activity scores: Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI)
Efficacy of the Treatment: BILAG | 5 years
  The change between baseline and post BAFF CAR-T cell infusion SLE disease activity scores: British Isles Lupus Assessment Group of SLE clinics (BILAG)
Efficacy of the Treatment: PGA | 5 years
  The change between baseline and post BAFF CAR-T cell infusion SLE disease activity scores: Physician Global Assessment (PGA) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Lee, PhD, Study Chair — Nationwide Children
Locations (1):
- Nationwide Children's, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No